CLINICAL TRIAL: NCT01239654
Title: Activity of Platelets After Inhibition and Cardiovascular Events: Drug Eluting Stent Implantation in Patients With Acute Coronary Syndrome: Optical Coherence Tomography Study
Brief Title: Activity of Platelets After Inhibition and Cardiovascular Events Optical Coherence Tomography Study
Acronym: APICE-OCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Mediolanum Cardio Research (Other); Cardiovascular Research Foundation, New York (Other)
Responsible Party: Principal Investigator, Antonio Colombo, Director of Invasive Cardiology, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APICE OCT Study (Project 4)
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Acute Coronary Syndrome
Keywords: acute; coronary; syndrome; everolimus; zotarolimus; optical; coherence; tomography
MeSH Terms: conditions — Acute Coronary Syndrome; Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- everolimus (Active Comparator): everolimus-eluting stent
  Interventions: Device: stent implantation
- zotarolimus (Active Comparator): zotarolimus-eluting stent
  Interventions: Device: stent implantation

INTERVENTIONS:
Device: stent implantation — implantation of everolimus-eluting stent vs zotarolimus-eluting stent

SUMMARY:
It is an exploratory study evaluating a biological effect (stent strut coverage) using a novel technology such as OCT without any clinical implication.

DETAILED DESCRIPTION:
The question of whether DES are safe, has become an area of considerable interest and controversy with the publication of a relatively small randomized trial (BASKET-LATE), an observational study and a meta-analysis reporting increased rates of ST, MI, and death with DES compared to BMS. The motivating factor was the presentation of a meta-analysis at the European Society of Cardiology meeting in Barcelona in September 2006, which suggested an increase in the risk of death and MI following implantation of sirolimus-eluting stents.

The major issue in these meta-analyses is that they were limited either by small sample sizes, duration of follow-ups, lack of access to source data, or by using landmark analyses that excluded events in first 6 months.

Moreover, the largest meta-analysis of DES vs. BMS and SES vs. PES published recently in The Lancet by Settler et al performed a network analyses with a mixed-treatment comparison of 38 randomized trials (18023 patients) with a follow-up of up to 4 years. This analysis again confirmed that DES and BMS were associated with similar rates of overall and cardiac mortality Regarding "real world" population, two observational registries recently published, i.e. the Western Denmark Heart Registry and the SCAAR (Swedish Coronary Angiography and Angioplasty Registry) confirmed no difference in the hard endpoints between DES and BMS. However, it must be remembered that these studies are observational and at best are hypothesis-generating.

Some autoptic studies have observed an incomplete healing following first generation DES implantation as compared to BMS; in these series late ST was associated with more delayed healing compared with patent DES. Among all the unsettled or not fully tested indications for usage of DES, ACS is most probably the one where implantation of BMS remains the most used approach because of the uncertainty regarding the thrombotic risk of DES in a thrombus rich milieu and the low risk for restenosis following BMS implantation in patients with acute MI. Despite encouraging results from currently published data with DES, well designed and appropriately powered clinical trials are warranted in order to establish long term safety and efficacy (incremental advantage over BMS) of DES in this setting. Moreover, recently it was reported that exposed struts were more frequent with first generation DES, and percent neointimal hyperplasia(NIH) area was smaller in ACS lesions than in non-ACS lesions.

For this specific purpose, we will evaluate, using OCT, complete neointimal coverage of Everolimus- vs. Zotarolimus Eluting Stent implanted in the novo lesions on native coronary arteries in patients with ACS. Rates of exposed and/or malaposed stent struts will be analysed and neointimal hyperplasia (NIH) area will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ACS and clinical indication to PCI
* Presence of 1 or more de novo stenosis equal or greater than 70% in native coronary arteries.
* Patient is > 18 years of age (or minimum age as required by local regulations).
* The patient has consented to participate by signing the "Patient Informed Consent Form".
* The patient is willing and able to cooperate with study procedures and required follow up visits.
* Any type of lesion can be included in this trial unless specifically detailed in the exclusion criteria.
* No other stent implanted before in the target lesion

Exclusion Criteria:

* Patients treated for lesions in venous or arterial grafts.
* Patients treated for in-stent restenosis.
* Patients treated for Unprotected Left Main lesions.
* Patients with left ventricular ejection fraction (LVEF) ≤30%.
* Patients with chronic kidney disease (creatinine ≥1.5 mg/dL) .
* Women with known pregnancy or who are lactating.
* Patients with hypersensitivity or allergies to heparin, drugs such as ABT-578 and everolimus, or any other analogue or derivative, cobalt, chromium, nickel, molybdenum or contrast media.
* Contraindication to the use of clopidogrel and/or ASA:

  1. History of drug allergy to thienopyridine derivatives or ASA;
  2. History of clinically significant or persistent thrombocytopenia or neutropenia
* Active bleeding or significant risk of bleedings, severe hepatic insufficiency, current peptic ulceration, proliferative diabetic retinopathy.
* Current medical condition with a life expectancy of less than 24 months.
* The subject is participating in another device or drug study. Subject must have completed the follow-up phase of any previous study at least 30 days prior to enrolment in this trial.
* Patients with medical conditions that preclude the follow-up as defined in the protocol or that otherwise limits participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the completeness of neointimal coverage following stent implantation (everolimus vs. zotarolimus-eluting stent) in patients with ACS. | 6 month
  Evaluate the completeness of neointimal coverage following stent implantation (everolimus vs. zotarolimus-eluting stent) in patients with ACS. The degree of neointimal coverage will be assessed using optical coherence tomography (OCT) calculating the rate of exposed stent struts in the study stents.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Colombo, MD, Principal Investigator — IRCCS San Raffaele
Locations (4):
- Italy (4):
  - Università della Magna Grecia, Catanzaro
  - Careggi Hospital, Florence
  - San Raffaele Hospital, Milan
  - Ospedale Civile di Mirano, Mirano

REFERENCES:
- [Background] Barlis P, Regar E, Serruys PW, Dimopoulos K, van der Giessen WJ, van Geuns RJ, Ferrante G, Wandel S, Windecker S, van Es GA, Eerdmans P, Juni P, di Mario C. An optical coherence tomography study of a biodegradable vs. durable polymer-coated limus-eluting stent: a LEADERS trial sub-study. Eur Heart J. 2010 Jan;31(2):165-76. doi: 10.1093/eurheartj/ehp480. Epub 2009 Nov 4. PMID 19889649
- [Background] Xie Y, Takano M, Murakami D, Yamamoto M, Okamatsu K, Inami S, Seimiya K, Ohba T, Seino Y, Mizuno K. Comparison of neointimal coverage by optical coherence tomography of a sirolimus-eluting stent versus a bare-metal stent three months after implantation. Am J Cardiol. 2008 Jul 1;102(1):27-31. doi: 10.1016/j.amjcard.2008.02.091. Epub 2008 Apr 25. PMID 18572031
- [Background] Matsumoto D, Shite J, Shinke T, Otake H, Tanino Y, Ogasawara D, Sawada T, Paredes OL, Hirata K, Yokoyama M. Neointimal coverage of sirolimus-eluting stents at 6-month follow-up: evaluated by optical coherence tomography. Eur Heart J. 2007 Apr;28(8):961-7. doi: 10.1093/eurheartj/ehl413. Epub 2006 Nov 29. PMID 17135281
- [Background] Tahara S, Bezerra HG, Sirbu V, Kyono H, Musumeci G, Rosenthal N, Guagliumi G, Costa MA. Angiographic, IVUS and OCT evaluation of the long-term impact of coronary disease severity at the site of overlapping drug-eluting and bare metal stents: a substudy of the ODESSA trial. Heart. 2010 Oct;96(19):1574-8. doi: 10.1136/hrt.2009.188037. Epub 2010 Aug 23. PMID 20736206
- [Background] Guagliumi G, Sirbu V, Bezerra H, Biondi-Zoccai G, Fiocca L, Musumeci G, Matiashvili A, Lortkipanidze N, Tahara S, Valsecchi O, Costa M. Strut coverage and vessel wall response to zotarolimus-eluting and bare-metal stents implanted in patients with ST-segment elevation myocardial infarction: the OCTAMI (Optical Coherence Tomography in Acute Myocardial Infarction) Study. JACC Cardiovasc Interv. 2010 Jun;3(6):680-7. doi: 10.1016/j.jcin.2010.04.005. PMID 20630463
- [Derived] Chieffo A, Buchanan GL, Parodi G, Versaci F, Bianchi RM, Valenti R, Sacca S, Mongiardo A, Span S, Migliorini A, Spaccarotella C, Reimers B, Antoniucci D, Indolfi C, Ferrari A, Maehara A, Mintz GS, Colombo A. Drug-eluting stent implantation in patients with acute coronary syndrome - the Activity of Platelets after Inhibition and Cardiovascular Events: Optical Coherence Tomography (APICE OCT) study. EuroIntervention. 2014 Dec;10(8):916-23. doi: 10.4244/EIJY14M06_10. PMID 24974806